CLINICAL TRIAL: NCT01827852
Title: AVAdeno: Non-interventional Study of Avastin 1st Line Therapy in Adenocarcinoma Patients of the Lung
Brief Title: AVAdeno Study: An Observational Study of First-Line Avastin (Bevacizumab) in Patients With Adenocarcinoma of the Lung
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28306
Record Dates: First submitted 2013-04-02; First posted 2013-04-10 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-06

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This prospective observational study will evaluate the efficacy and safety of first-line Avastin (bevacizumab) in combination with platinum-based chemotherapy in different age groups (<60, 60-69, 70-79, >80 years) in patients with inoperable advanced, metastatic or recurrent adenocarcinoma non-small cell lung cancer. Patients will be followed for 18 months from the start of first-line therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Histologically confirmed inoperable advanced, metastatic or recurrent pre-dominantly non-squamous adenocarcinoma non-small cell lung cancer

Exclusion Criteria:

* Contraindications to Avastin treatment according to the Summary of Product Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with inoperable advanced, metastatic or recurrent predominantly non-squamous adenocarcinoma non-small cell lung cancer
Sampling Method: Probability Sample
Enrollment: 1107 (Actual)
Dates: Start 2013-03-14 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Progression-free survival in 4 different age groups (<60, 60-69, 70-79, >/=80 years) | approximately 4.5 years

SECONDARY OUTCOMES:
Overall survival in 4 different age groups (<60, 60-69, 70-79, >/=80 years) | approximately 4.5 years
Clinical/demographic patient characteristics at initiation of treatment | approximately 4.5 years
Avastin treatment schedule in routine clinical practice (dosage/duration) | approximately 4 years
Concomitant anti-neoplastic therapy (dosage/duration) | approximately 4.5 years
Safety: Incidence of adverse events in 4 different age groups (<60, 60-69, 70-79, >/=80 years) | approximately 4.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Universität Leipzig; Medizinische Klinik und Poliklinik I, Abteilung Pneumologie, Leipzig, Germany